CLINICAL TRIAL: NCT04946253
Title: Care Team and Practice Level Implementation Strategies to Optimize Pediatric Collaborative Care: A Cluster-Randomized Trial
Brief Title: SKIP for PA Study: Team and Leadership Level Implementation Support for Collaborative Care
Acronym: SKIPforPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Academy of Pediatrics (Other); Drexel University (Other); NYU Langone Health (Other); University of Michigan (Other); National Institute of Mental Health (NIMH) (NIH); Pennsylvania American Academy of Pediatrics (Unknown)
Responsible Party: Principal Investigator, David Kolko, Professor of Psychiatry, Psychology, Pediatrics, and Clinical and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20080207; R01MH124914 (NIH)
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Child Behavior Problem; Attention Deficit and Disruptive Behavior Disorders
Keywords: Oppositional Defiant Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The investigators propose a randomized trial using a factorial design to test effects of implementation support strategies on uptake of an evidence-based intervention (DOCC) in up to 24 primary care practices. Practices will receive DOCC training in accord with the Replicating Effective Programs model. Practices will be randomized to 1 of 4 implementation support conditions: 1) No TEAM/LEAD (training and technical support only); 2) provider care team consultation (TEAM); 3) practice leadership facilitation (LEAD); and 4) combination of provider care team and leadership implementation (TEAM+LEAD). Care teams in each practice will identify families and deliver DOCC to 20 caregivers and their children with externalizing behavior. Investigators will collect measures from 90 practice staff over 5 assessments (24 months) and 360 caregivers over 4 assessments (12 months) to support analyses.
Who Masked: Outcomes Assessor
Masking Description: Participants are not directly informed of the implementation condition to which the practice site has been randomized. All formal standardized assessments will be conducted via secure electronic web-based data collection systems, limiting the potential for assessment bias. In the event that a caregiver requests that a staff member administer an assessment via phone, the assessor would be unaware of the implementation condition assigned to the child's practice where the caregiver receives care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DOCC with standard implementation (No TEAM or LEAD) (Active Comparator): Practices in this arm will receive DOCC materials/training and technical support, but will not receive care team coaching/consultation (TEAM) or practice leadership facilitation (LEAD) after the training phase.
  Interventions: Behavioral: DOCC: Evidence-based treatment for disruptive behavior and ADHD
- DOCC with TEAM implementation (Experimental): Practices in this arm will receive DOCC training and materials and one type of implementation support after the training: coaching/consultation for the provider care team (TEAM).
  Interventions: Behavioral: DOCC: Evidence-based treatment for disruptive behavior and ADHD; Behavioral: TEAM: Implementation support strategies at the care team level following standard implementation of DOCC
- DOCC with LEAD implementation (Experimental): Practices in this arm will receive DOCC training and materials and only one type of implementation support after the training: facilitation for practice leadership (LEAD).
  Interventions: Behavioral: DOCC: Evidence-based treatment for disruptive behavior and ADHD; Behavioral: Implementation support strategies at the leadership level following standard implementation of DOCC
- DOCC with TEAM + LEAD implementation (Experimental): Practices in this arm will receive DOCC training and materials and both types of implementation support after the training: coaching/consultation for the provider care team (TEAM) and facilitation for practice leadership (LEAD).
  Interventions: Behavioral: DOCC: Evidence-based treatment for disruptive behavior and ADHD; Behavioral: TEAM: Implementation support strategies at the care team level following standard implementation of DOCC; Behavioral: Implementation support strategies at the leadership level following standard implementation of DOCC

INTERVENTIONS:
Behavioral: DOCC: Evidence-based treatment for disruptive behavior and ADHD — Practices will learn and then deliver DOCC in treatment sessions with caregivers and/or children. The content covers key topics related to the treatment of behavior problems (e.g., self-management, positive parenting) and ADHD (e.g., psychoeducation, medication).
Behavioral: TEAM: Implementation support strategies at the care team level following standard implementation of DOCC — Practices will learn and then deliver DOCC in treatment sessions with caregivers and/or children. Coaching and consultation will be provided to the provider care team to support the use of collaborative care for behavior problems and ADHD. The TEAM intervention includes regular virtual meetings or calls with the providers (about once/month, on average) that cover core chronic care model functions, including registry use, case-finding, collaborative care team roles, and workflows outlining how DOCC is delivered in the practice.
  Arms: DOCC with TEAM + LEAD implementation; DOCC with TEAM implementation
Behavioral: Implementation support strategies at the leadership level following standard implementation of DOCC — Practices will learn and then deliver DOCC in treatment sessions with caregivers and/or children. Practice facilitation will be provided to practice leaders to help them support the care team's use of collaborative care for behavior problems and ADHD. The LEAD intervention includes regular virtual meetings or calls with practice leaders (about once/month, on average) that cover the assessment of practice capacity/barriers, ways to overcome organizational barriers and support staff use of DOCC, promoting innovation, and leveraging practice resources to support DOCC delivery and maintenance in the practice.
  Arms: DOCC with LEAD implementation; DOCC with TEAM + LEAD implementation

SUMMARY:
In a prior application (MH064372), the investigators' treatment research program (Services for Kids In Primary-care, SKIP) developed and tested a chronic care model-based intervention, called Doctor Office Collaborative Care (DOCC), that was found to be effective in the management of childhood behavior problems and comorbid ADHD. In the "SKIP for PA Study", the investigators propose to conduct a randomized clinical trial to evaluate the effects of team- and practice leadership-level implementation strategies designed to enhance the use and uptake of DOCC in diverse pediatric primary care offices.

DETAILED DESCRIPTION:
This study is a randomized, hybrid type 3 effectiveness-implementation trial to support the adoption of a chronic care model (CCM)-based intervention in pediatric primary care settings by testing the impact of implementation strategies directed towards the provider care team (TEAM) or practice leadership (LEAD) level. The treatment investigators seek to deliver here is called Doctor Office Collaborative Care (DOCC), an evidence-based intervention for the management of child behavior problems and comorbid ADHD. The implementation strategies being tested to enhance DOCC uptake include TEAM coaching/consultation strategies, which will be delivered to care team providers and target provider competency to deliver DOCC, and LEAD facilitation strategies, which will be delivered to practice leaders and target organizational support of DOCC delivery. These multi-level implementation strategies have not been formally evaluated to learn about their separate and combined effects in any randomized clinical trial conducted in pediatric primary care. Such information is needed to optimize our approaches to promoting the implementation of a CCM-based intervention in pediatric practice.

The sample includes up to 24 primary care practices from a statewide network and other networks or states. After standard training in the DOCC EBP, all practices will be randomized to one of four implementation conditions: 1) No TEAM or LEAD (ongoing technical support only); 2) TEAM implementation; 3) LEAD implementation, or 4) TEAM+LEAD implementation. TEAM and LEAD implementation will be delivered via videoconference on a graded schedule. Care teams will deliver DOCC to up to 25 children (or more if requested by the practice) who meet a clinical cutoff for modest behavior problems and their caregivers. Investigators will collect practice/provider measures from enrolled practice staff (0, 6, 12, 18, 24 months) and caregivers over several timepoints (0, 3, 6, 12 months) to support all analyses evaluating implementation and treatment outcomes, mediation, and moderation. By proposing one of the first large pragmatic pediatric trials of a CCM-based evidence-based intervention to address these aims in response to RFA-MH-18-701 and the NIMH's Strategic Plan (4.2), this research will advance the implementation science knowledge needed to optimize promising strategies for promoting the delivery and scale-up of DOCC in a pediatric medical home.

ELIGIBILITY:
The investigators propose to recruit 4 types of practice provider participants (PCP = primary care provider, CM = care manager, SL = Senior Leader, PM = practice manager) as well as caregiver participants.

Inclusion Criteria:

* PCP Participants:

  * Employed at one of the up to twenty-four (24) pediatric primary care practices identified by the PA Medical Home Program at the PA AAP or by the University of Pittsburgh research team.
  * Identified by the practice as a Primary Care Provider
* CM Participants:

  * Employed at one of the up to twenty-four (24) pediatric primary care practices identified by the PA Medical Home Program at the PA AAP or by the University of Pittsburgh research team.
  * Identified by the practice as a Behavioral Health Resource who delivers and coordinates behavioral health care in the practice, who will function in the study as a care manager.
* SL Participants:

  * Employed at one of the up to twenty-four (24) pediatric primary care practices identified by the PA Medical Home Program at the PA AAP or by the University of Pittsburgh research team.
  * Identified by the practice as the Senior Leader.
  * Have a practice-level leadership role such as Medical Director or a clinical/practice leader
  * Have administrative responsibilities related to patient care and/or the operations/management of the practice
* PM Participants:

  * Employed at one of the up to twenty-four (24) pediatric primary care practices identified by the PA Medical Home Program at the PA AAP or by the University of Pittsburgh research team.
  * Identified by the practice as the Practice Manager or equivalent position
  * Are responsible for day-to-day practice operations, such as personnel management, billing, and compliance with regulations, in the pediatric practice.
* Caregiver Participants:

  * Have a child age 5-12 years old who exhibits at least a modest level of behavior problems (Caregiver Participants)
  * Are at least 18 years of age (Caregiver participants)
  * Have parental rights for this child (Caregiver participants)

Exclusion Criteria:

* Caregivers

  * Already enrolled in the study as the caregiver to a different child (e.g., sibling) (Caregiver participants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Total number of DOCC encounters | Throughout services after each contact, up to 12 months
  As part of a short checklist-style progress note completed after each service contact and housed in the study's web-based patient registry dashboard, providers will document each DOCC encounter delivered to each family. These encounters include referral, assessment, treatment or medication delivery, medication or treatment review/monitoring, case management, review of emergent symptoms, and care management and consultation meetings involving a family member. Investigators will report the total number of DOCC encounters delivered to each family during the intervention phase.
Care management competencies and functions | At provider baseline
  The Mental Health Practice Readiness Inventory will be completed to document the degree to which a practice has the organizational and individual competencies needed to support integrated BH care. All 32 items reflect the diverse activities (e.g., workflows, financing, service delivery, care coordination) suggested as functions for PCPs (scale: 0 = no function exists; 1 = some function; 2 = function is complete). Thus, total scale scores can range from 0 to 64. Investigators will use scores for each of the 32 competency items (range 0-2) and the total score (range 0-64) to describe the overall level of collaborative care competencies achieved per practice.
Change from baseline in care management competencies and functions at 6 months | 6 months after provider baseline
  The Mental Health Practice Readiness Inventory will be completed to document the degree to which a practice has the organizational and individual competencies needed to support integrated BH care. All 32 items reflect the diverse activities (e.g., workflows, financing, service delivery, care coordination) suggested as functions for PCPs (scale: 0 = no function exists; 1 = some function; 2 = function is complete). Thus, total scale scores can range from 0 to 64. Investigators will use scores for each of the 32 competency items (range 0-2) and the total score (range 0-64) to describe the overall level of collaborative care competencies achieved per practice.
Change from baseline in care management competencies and functions at 12 months | 12 months after provider baseline
  The Mental Health Practice Readiness Inventory will be completed to document the degree to which a practice has the organizational and individual competencies needed to support integrated BH care. All 32 items reflect the diverse activities (e.g., workflows, financing, service delivery, care coordination) suggested as functions for PCPs (scale: 0 = no function exists; 1 = some function; 2 = function is complete). Thus, total scale scores can range from 0 to 64. Investigators will use scores for each of the 32 competency items (range 0-2) and the total score (range 0-64) to describe the overall level of collaborative care competencies achieved per practice.
Change from baseline in care management competencies and functions at 18 months | 18 months after provider baseline
  The Mental Health Practice Readiness Inventory will be completed to document the degree to which a practice has the organizational and individual competencies needed to support integrated BH care. All 32 items reflect the diverse activities (e.g., workflows, financing, service delivery, care coordination) suggested as functions for PCPs (scale: 0 = no function exists; 1 = some function; 2 = function is complete). Thus, total scale scores can range from 0 to 64. Investigators will use scores for each of the 32 competency items (range 0-2) and the total score (range 0-64) to describe the overall level of collaborative care competencies achieved per practice.
Change from baseline in care management competencies and functions at 24 months | 24 months after provider baseline
  The Mental Health Practice Readiness Inventory will be completed to document the degree to which a practice has the organizational and individual competencies needed to support integrated BH care. All 32 items reflect the diverse activities (e.g., workflows, financing, service delivery, care coordination) suggested as functions for PCPs (scale: 0 = no function exists; 1 = some function; 2 = function is complete). Thus, total scale scores can range from 0 to 64. Investigators will use scores for each of the 32 competency items (range 0-2) and the total score (range 0-64) to describe the overall level of collaborative care competencies achieved per practice.
Severity of ADHD, ODD, CD, and ANX/DEP symptoms at home and in community | At caregiver baseline
  To assess the severity of the child's behavioral and emotional problems, the Vanderbilt ADHD Diagnostic Rating Scale will be completed by caregivers. The VADPRS includes 5 symptom severity subscales, each with a varying number of items: (hyperactivity/impulsivity (n=9), inattention (n=9), oppositional behavior (n=7), conduct problems (n=15), and anxiety/depression (n=7). The scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance (impairment) subscale (n=7) used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional behavior (21), conduct problems (45), anxiety/depression (21) ,and performance (24).
Change from baseline in severity of ADHD, ODD, CD, and ANX/DEP symptoms at home and in community at 3 months | 3 months after caregiver baseline
  To assess the severity of the child's behavioral and emotional problems, the Vanderbilt ADHD Diagnostic Rating Scale will be completed by caregivers. The VADPRS includes 5 symptom severity subscales, each with a varying number of items: (hyperactivity/impulsivity (n=9), inattention (n=9), oppositional behavior (n=7), conduct problems (n=15), and anxiety/depression (n=7). The scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance (impairment) subscale (n=7) used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional behavior (21), conduct problems (45), anxiety/depression (21) ,and performance (24).
Change from baseline in severity of ADHD, ODD, CD, and ANX/DEP symptoms at home and in community at 6 months | 6 months after caregiver baseline
  To assess the severity of the child's behavioral and emotional problems, the Vanderbilt ADHD Diagnostic Rating Scale will be completed by caregivers. The VADPRS includes 5 symptom severity subscales, each with a varying number of items: (hyperactivity/impulsivity (n=9), inattention (n=9), oppositional behavior (n=7), conduct problems (n=15), and anxiety/depression (n=7). The scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance (impairment) subscale (n=7) used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional behavior (21), conduct problems (45), anxiety/depression (21) ,and performance (24).
Change from baseline in severity of ADHD, ODD, CD, and ANX/DEP symptoms at home and in community at 12 months | 12 months after caregiver baseline
  To assess the severity of the child's behavioral and emotional problems, the Vanderbilt ADHD Diagnostic Rating Scale will be completed by caregivers. The VADPRS includes 5 symptom severity subscales, each with a varying number of items: (hyperactivity/impulsivity (n=9), inattention (n=9), oppositional behavior (n=7), conduct problems (n=15), and anxiety/depression (n=7). The scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance (impairment) subscale (n=7) used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional behavior (21), conduct problems (45), anxiety/depression (21) ,and performance (24).
Severity of ADHD, ODD/CD, and ANX/DEP symptoms at school | At teacher baseline
  Paralleling the VADPRS, the VADTRS will be completed by teachers. This version includes 3 of the same subscales in the parent version -- hyperactivity/impulsivity (n=9), inattention (n=9), and anxiety/depression (n=7) -- but it also includes an aggregated oppositional/conduct scale (n=10 items). Scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance subscale (n=8 items) that is used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional/conduct problems (30), anxiety/depression (21) ,and performance (24). Practices will continue to separately request their own forms during services (e.g., for medication monitoring).
Change from baseline in severity of ADHD, ODD/CD, and ANX/DEP symptoms at school at 3 months | 3 months after teacher baseline
  Paralleling the VADPRS, the VADTRS will be completed by teachers. This version includes 3 of the same subscales in the parent version -- hyperactivity/impulsivity (n=9), inattention (n=9), and anxiety/depression (n=7) -- but it also includes an aggregated oppositional/conduct scale (n=10 items). Scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance subscale (n=8 items) that is used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional/conduct problems (30), anxiety/depression (21) ,and performance (24). Practices will continue to separately request their own forms during services (e.g., for medication monitoring).
Change from baseline in severity of ADHD, ODD/CD, and ANX/DEP symptoms at school at 6 months | 6 months after teacher baseline
  Paralleling the VADPRS, the VADTRS will be completed by teachers. This version includes 3 of the same subscales in the parent version -- hyperactivity/impulsivity (n=9), inattention (n=9), and anxiety/depression (n=7) -- but it also includes an aggregated oppositional/conduct scale (n=10 items). Scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance subscale (n=8 items) that is used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional/conduct problems (30), anxiety/depression (21) ,and performance (24). Practices will continue to separately request their own forms during services (e.g., for medication monitoring).
Change from baseline in severity of ADHD, ODD/CD, and ANX/DEP symptoms at school at 12 months | 12 months after teacher baseline
  Paralleling the VADPRS, the VADTRS will be completed by teachers. This version includes 3 of the same subscales in the parent version -- hyperactivity/impulsivity (n=9), inattention (n=9), and anxiety/depression (n=7) -- but it also includes an aggregated oppositional/conduct scale (n=10 items). Scores for the hyperactivity/impulsivity and inattention subscales are often aggregated to create an overall ADHD scale factor total score. Individual items are rated on a 4-point Likert scale (0 = never; 1 = occasionally; 2 = often; 3 = very often). There is also a performance subscale (n=8 items) that is used to determine whether a child would meet clinical criteria for a given disorder. The range of scores per factor are as follows: hyperactivity/impulsivity (27), inattention (27), oppositional/conduct problems (30), anxiety/depression (21) ,and performance (24). Practices will continue to separately request their own forms during services (e.g., for medication monitoring).
Pediatric Health Quality | At caregiver baseline
  Caregivers will complete the Pediatric Quality of Life (PEDS-QL) to measure health-related quality of life which includes 4 subscales: health/physical status (n=8), emotional health (n=5), school health (n=5), and social health (n=5). All items are rated on a 5-point Likert scale (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). These subscales have very good reliability and treatment validity and are sensitive to the DOCC EBP.
Change from baseline in Pediatric Health Quality at 3 months | 3 months after caregiver baseline
  Caregivers will complete the Pediatric Quality of Life (PEDS-QL) to measure health-related quality of life which includes 4 subscales: health/physical status (n=8), emotional health (n=5), school health (n=5), and social health (n=5). All items are rated on a 5-point Likert scale (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). These subscales have very good reliability and treatment validity and are sensitive to the DOCC EBP.
Change from baseline in Pediatric Health Quality at 3 months | 6 months after caregiver baseline
  Caregivers will complete the Pediatric Quality of Life (PEDS-QL) to measure health-related quality of life which includes 4 subscales: health/physical status (n=8), emotional health (n=5), school health (n=5), and social health (n=5). All items are rated on a 5-point Likert scale (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). These subscales have very good reliability and treatment validity and are sensitive to the DOCC EBP.
Change from baseline in Pediatric Health Quality at 12 months | 12 months after caregiver baseline
  Caregivers will complete the Pediatric Quality of Life (PEDS-QL) to measure health-related quality of life which includes 4 subscales: health/physical status (n=8), emotional health (n=5), school health (n=5), and social health (n=5). All items are rated on a 5-point Likert scale (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). These subscales have very good reliability and treatment validity and are sensitive to the DOCC EBP.
Professional perceptions of study experiences at 18 months | 18 months after professional baseline
  Professionals will be invited to participate in an 18-month qualitative interview after they complete their 18-month online assessment. The purpose of this research interview is to provide feedback about their experiences with different aspects of this study, such as: learning and using the DOCC intervention, working as a team, participating any facilitation calls, and completing our research tasks. The interview gives us unique information about their perspective on these topics that can help us extend what we can learn from their surveys and then modify or tailor any of these methods to better support feasibility and acceptability. All responses will be thematically coded and summarized for interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: David J Kolko, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case data, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. Study investigators/study staff will upload descriptive/raw data to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis. Data will be released to NDCT after manuscripts reporting primary findings are accepted for publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication. The investigators plan to make these data available indefinitely, with no anticipated time limit.
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting the principal investigator.

REFERENCES:
- [Background] Dikhanov GG, Mishan'kin BN. [Comparative study of ribosomal proteins from Yersinia pestis and Escherichia coli: amino acid composition and electrophoretic mobility]. Mol Gen Mikrobiol Virusol. 1988 Aug;(8):32-5. Russian. PMID 3057358
- [Background] Kolko DJ, Campo JV, Kilbourne AM, Kelleher K. Doctor-office collaborative care for pediatric behavioral problems: a preliminary clinical trial. Arch Pediatr Adolesc Med. 2012 Mar;166(3):224-31. doi: 10.1001/archpediatrics.2011.201. Epub 2011 Nov 7. PMID 22064876
- [Background] Tsai CC, Williamson HO, Kirkland BH, Braun JO, Lam CF. Low-dose oral contraception and blood pressure in women with a past history of elevated blood pressure. Am J Obstet Gynecol. 1985 Jan 1;151(1):28-32. doi: 10.1016/0002-9378(85)90418-1. PMID 3966503
- [Background] Ballogh Z, Whaley K. Hereditary angio-oedema: its pathogenesis and management. Scott Med J. 1980 Jul;25(3):187-95. doi: 10.1177/003693308002500303. PMID 7444430
- [Background] McGuier EA, Kolko DJ, Ramsook KA, Huh AS, Berkout OV, Campo JV. Effects of Primary Care Provider Characteristics on Changes in Behavioral Health Delivery During a Collaborative Care Trial. Acad Pediatr. 2020 Apr;20(3):399-404. doi: 10.1016/j.acap.2019.11.008. Epub 2019 Nov 21. PMID 31760174
- [Background] Glukhen'kii TT, Gude ZZh. [The blood level of certain monosaccharides in patients with eczema]. Vestn Dermatol Venerol. 1969 Apr;43(4):33-5. No abstract available. Russian. PMID 5364816
- [Background] Paoni NF, Keyt BA, Refino CJ, Chow AM, Nguyen HV, Berleau LT, Badillo J, Pena LC, Brady K, Wurm FM, et al. A slow clearing, fibrin-specific, PAI-1 resistant variant of t-PA (T103N, KHRR 296-299 AAAA). Thromb Haemost. 1993 Aug 2;70(2):307-12. PMID 8236140
- [Background] Meier DA, Nagle CE. Differential diagnosis of a tender goiter. J Nucl Med. 1996 Oct;37(10):1745-7. PMID 8862323
- [Derived] Kolko DJ, McGuier EA, Turchi R, Thompson E, Iyengar S, Smith SN, Hoagwood K, Liebrecht C, Bennett IM, Powell BJ, Kelleher K, Silva M, Kilbourne AM. Care team and practice-level implementation strategies to optimize pediatric collaborative care: study protocol for a cluster-randomized hybrid type III trial. Implement Sci. 2022 Feb 22;17(1):20. doi: 10.1186/s13012-022-01195-7. PMID 35193619